CLINICAL TRIAL: NCT01959386
Title: Clinical Practice Surveillance of the Use of Herceptin® Subcutaneous in Patients With HER2-Positive Early Breast Cancer (HerSCin)
Brief Title: A Study of Trastuzumab Subcutaneous in Participants With Human Epidermal Growth Factor Receptor-2 (HER2) Positive Early Breast Cancer
Acronym: HerSCin
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28759
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2 Positive Breast Cancer Participants: Participants with HER2 positive tumors who are considered for treatment with trastuzumab SC according to the judgement of physician and according to the actual summary of product characteristics will be observed for a period of approximately 1 year and will be followed for an additional 2 years.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Participants will be receiving trastuzumab as part of their treatment for breast cancer according to the judgement of physician and according to the actual summary of product characteristics. The study protocol does not influence the physician's decision regarding diagnostics, therapy or frequency of medical examination during or after the treatment.
  Other Names: Herceptin

SUMMARY:
This observational study will evaluate the efficacy, safety, tolerability and participant reported quality of life of trastuzumab (Herceptin) subcutaneous (SC) therapy in participants with HER2-positive early breast cancer in routine clinical practice. Data from eligible participants will be collected for the duration of their treatment (approximately 1 year) and for 1-2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast
* HER2-positive tumor
* Eligible for neo-adjuvant or adjuvant treatment with trastuzumab SC according to the judgement of the physician Note: As of participant recruitment (date of participant informed consent), retrospective documentation is allowed but limited to up to 9 weeks after initial start of therapy with trastuzumab SC

Exclusion Criteria:

* Contraindications according to the Summary of Product Characteristics of Herceptin SC
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HER2-positive early breast cancer initiated on treatment with subcutaneously administered trastuzumab.
Sampling Method: Non-Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Pathologic Complete Response (pCR) (For Participants Treated in Neo-Adjuvant Setting), According to Response Evaluation Criteria in Solid Tumor (RECIST), or Modified RECIST, or Cheson Criteria (As per Center Practice) | Baseline up to approximately 3 years (assessed according to routine center practice)
Percentage of Participants Who Were Alive and Disease Free at Year 2 (For Participants Treated in the Adjuvant Setting), According to RECIST, or Modified RECIST, or Cheson Criteria (As per Center Practice) | Year 2

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to approximately 3 years
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) Scores | Baseline, every 12 weeks up to Year 1
European Organization for Research and Treatment of Cancer Breast Cancer Module (EORTC QLQ BR23) Questionnaire Score | Baseline, every 12 weeks up to Year 1
Mean Trastuzumab Dose | Baseline up to Year 1
Duration of Trastuzumab Treatment | Baseline up to Year 1
Percentage of Participants By Reason for Trastuzumab Discontinuation or Interruption | Baseline up to Year 1
Percentage of Participants Who Received Concomitant Treatment (Chemotherapy or Any Other Treatment) | Baseline up to Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz, Germany